CLINICAL TRIAL: NCT02267915
Title: An Open Multicenter Phase II Study of Efficacy and Toxicity of Maintenance Subcut. Rituximab After Induction With Rituximab in Patients With Relapsed or Refractory Mantle-cell Lymphoma Non-eligible for HSCT
Brief Title: Phase II of Efficacy and Toxicity of Maintenance Sub. Rituximab After Induction in Relapsed MCL and Non-eligible HSCT
Acronym: MAN2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Grupo Español de Linfomas y Transplante Autólogo de Médula Ósea (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GELTAMO-MAN2
Record Dates: First submitted 2014-10-03; First posted 2014-10-20 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2019-05

CONDITIONS: Mantle-cell Lymphoma
Keywords: Relapsed or refractory patients with mantle-cell lymphoma; Progression after high-dose chemotherapy and autologous HPT
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Recurrence | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- subcutaneous rituximab (Experimental): MabThera 1400 mg solution for subcutaneous injection
  Interventions: Drug: subcutaneous Rituximab

INTERVENTIONS:
Drug: subcutaneous Rituximab — MabThera 1400 mg solution for subcutaneous injection
  Other Names: MABTHERA

SUMMARY:
1. Primary endpoint: Time to relapse/progression (TTP) after achieving a complete or partial response with the (R-GemOxD)-induction therapy
2. Secondary endpoints:

   1. Quality of response obtained after subcutaneous Rituximab maintenance.
   2. Progression-Free Survival (PFS)
   3. Overall Survival (OS)
   4. Time to Next Therapy (TTNT)
   5. Value of MRD in the disease outcome
   6. Toxicity

DETAILED DESCRIPTION:
This is a phase II trial evaluating the role of maintenance with subcutaneous Rituximab in patients with stage II-IV relapsed or refractory mantle-cell lymphoma with complete or partial response after the administration of a salvage regimen with R-GemOx-D.

Before the study start and in order to standardize the results, the same R-GemOx-D salvage regimen will be used: Rituximab: 375 mg/m2 on day 1, Gemcitabine: 1000 mg/m2 on day 2 (over 30 minutes) and Oxaliplatin: 100 mg/m2 on day 2 (over 3 hours), Dexamethasone 20 mg on day 1-3. Cycles should be repeated every 14 days, up to 8 cycles.

Patients who present a complete or partial response, after the salvage therapy, will start the study receiving subcutaneous Rituximab maintenance at dose of: 1400 mg every 2 months for 2 years; the study treatment will start 6-8 weeks after finishing the salvage therapy.

Patients will be evaluated every 2 months during treatment study phase and every 4 months in the follow up phase. More details in Appendix 1 (Schedule of Assessments)

ELIGIBILITY:
Inclusion Criteria:

* Basal diagnosis of mantle-cell lymphoma in relapse or refractory.
* Achievement of a CR or PR after salvage therapy with R-GemOxD (6 to 8 cycles) as previously described4-5.
* Age > 18 years.
* One or maximum two prior chemotherapy or immunochemotherapy lines.
* Patients should not be considered candidates for high-dose chemotherapy and autologous stem-cell transplantation.
* No clinical evidence of CNS involvement
* Signed informed consent
* Serum creatinine less than 2 and/or bilirrubin less than 2.5 UNL.
* Pregnant or lactating woman. FCBP must agree to ongoing pregnancy testing during the course or study and commit to use effective contraception during the study

Exclusion Criteria:

* Prior organ transplantation.
* HIV positive.
* HBV related disease
* Any serious active disease or co-morbid medical condition (according to the investigator's decision)
* Any history of cancer during the last 5 years, with the exception of non-melanoma skin tumors or stage 0 cervix carcinoma.
* Less than 50% of tumor response.
* Platelet counts less than 50 x 109/L.
* Neutrophil counts less than 1.0 x 109/L.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2015-03 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Time to progression, (Measured from achievement of response -partial or complete- to to disease progression) | 2 YEARS
  2 years after last patient randomized in maintenance

CONTACTS AND LOCATIONS:
Overall Officials: Andres Lopez, DOCTOR, Study Director — Grupo Español de Linfomas y Transplante Autólogo de Médula Ósea
Locations (11):
- Spain (11):
  - Geltamo Investigational Site, Santiago de Compostela, LA Coruña
  - Geltamo Investigational Site, Alcorcón, Madrid
  - Geltamo Investigational Site, Majadahonda, Madrid
  - Geltamo Investigational Site, Gijón, Principality of Asturias
  - Geltamo Investigational Site, Barcelona
  - Geltamo Investigational Site, Burgos
  - Geltamo Investigational Site, Granada
  - Geltamo Investigational Site, Madrid
  - Geltamo Investigational Site, Salamanca
  - Geltamo Investigational Site, Santander
  - Geltamo Investigational Site, Seville